CLINICAL TRIAL: NCT02704689
Title: A Prospective Multi-Center Evaluation of a Hydraulic Expandable TLIF Cage for the Treatment of Degenerative Disc Disease of the Lumbar Spine
Brief Title: AccuLIF® PROSPECTIVE PATIENT OUTCOMES STUDY
Acronym: APROPOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment
Sponsor: Stryker Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-L-001; 510(k) 132505 & K143616 (Other: U.S. Food and Drug Administration)
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis, Grade 1; Retrolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AccuLIF (Experimental)
  Interventions: Device: AccuLIF expandable TLIF cage

INTERVENTIONS:
Device: AccuLIF expandable TLIF cage — AccuLIF TL expandable interbody cage used with autogenous bone and/or allograft (cancellous or corticocancellous allograft chips) and supplemental fixation.

SUMMARY:
This is a post-market clinical study of the AccuLIF expandable transforaminal lumbar interbody fusion (TLIF) cage in patients requiring surgery for degenerative disc disease (DDD) with up to Grade I spondylolisthesis or retrolisthesis, at one or two levels, between L2 and S1.

DETAILED DESCRIPTION:
Study evaluations will be evaluated pre-operatively and at 6-weeks, 3-months, 6-months, 12-months and 24-months post-operatively to assess clinical outcomes, patient reported outcomes and radiographic status.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is skeletally mature and between 18 and 70 years of age.
2. DDD and up to Grade I spondylolisthesis or retrolisthesis, requiring decompression and arthrodesis at one or two contiguous levels between L2 and S1.
3. No previous surgery at the same or adjacent level (other than microdiscectomy / laminectomy) at the same or adjacent level.
4. Non-responsive to conservative (non-surgical) treatment for back pain for a minimum of 6 months.
5. Subject understands the conditions of enrollment and is willing to sign and date the Informed Consent.
6. Subject agrees to comply with visit schedule and completing study questionnaires.

Exclusion Criteria:

1. Significant instability of the spine.
2. Requires TLIF at more than 2 levels between L2 and S1.
3. Previously undergone lumbar spine surgery (other than microdiscectomy / laminectomy) at the same or adjacent level.
4. Younger than 18 years of age, or older than 70 years of age.
5. BMI of 40 or greater.
6. History of metabolic bone disease
7. Osteoporosis
8. Diabetes mellitus requiring daily insulin management.
9. Subject has any of the following:

   1. Progressive neuromuscular disease; OR
   2. Autoimmune disease; OR
   3. Active malignancy within the last 15 years; OR
   4. Active hepatitis; OR
   5. AIDS, ARC, or is HIV positive; OR
   6. Syringomyelia at any spinal level; OR
   7. Any other condition that would interfere with the subject self -assessment of pain, function or quality of life.
10. Allergy to implant materials (titanium, titanium alloy).
11. Active systemic infection or infection localized to the site of implantation.
12. Primary or metastatic tumors involving the spine.
13. Open wounds or inadequate issue tissue coverage over the operative site.
14. History of significant mental illness or mental incapacity.
15. Pregnancy or intent to become pregnant.
16. Participating in another investigational study for a similar purpose.
17. Belongs to a vulnerable population that would compromise ability to provide informed consent or compliance with follow-up requirements.
18. Smokers unwilling to cease up to 3 months post-op or recent history of alcohol or other substance abuse within the past 2 years.
19. Workers compensation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Choma, MD, Principal Investigator — University of Missouri Health Care
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AccuLIF TL: All subjects enrolled were assigned to receive lumbar interbody fusion via a TLIF approach with the AccuLIF TL cage.
Period: Overall Study
Arm/Group | AccuLIF TL
Started | 9
Completed | 6
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Study device not implanted | 2

BASELINE CHARACTERISTICS:
Population: Total enrollment
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 32 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Radiographic Measurements to Evaluate Segmental Lordosis as Measured by Degree of Change From Pre-operative X-rays.
Description: Post-operative radiographic measurements to evaluate segmental lordosis as measured by degree of change from pre-operative x-rays.
Time Frame: 24 months
Population: The Primary Outcome Measures were going to be analyzed at the 24 month visit. However, this study was terminated early due to lack of enrollment and no subjects reached the 24 month analysis visit. There is, therefore, no data to summarize for this Primary Outcome Measure.
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

2. Primary Outcome: Pre-operative Comparison to Post-operative Radiographic Outcomes of Disc Height as Measured in mm.
Description: Pre-operative comparison to post-operative radiographic outcomes of disc height as measured in mm.
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

3. Secondary Outcome: Surgical Outcomes: To Measure the Length of Surgery as Measured in Time of Surgery Duration.
Description: Surgical Outcomes: To measure the length of surgery as measured in time of surgery duration.
Time Frame: Operative Visit
Population: Subjects treated with the AccuLIF TL device
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 6
minutes | 192 (35)

4. Secondary Outcome: Surgical Outcomes: To Evaluate the Length of Time Hospitalized for the Index Procedure as Measured in Days.
Description: Surgical Outcomes: To evaluate the length of time hospitalized for the index procedure as measured in days.
Time Frame: Peri-op
Population: Subjects treated with the AccuLIF TL device
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 6
days | 4 (2.7)

5. Secondary Outcome: Surgical Outcomes: To Measure the Amount of Blood Loss at the Time of Surgery.
Description: Surgical Outcomes: To measure the amount of blood loss at the time of surgery.
Time Frame: Operative Visit
Population: Subjects treated with the AccuLIF TL device
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 6
cc | 383 (311)

6. Secondary Outcome: Medical Outcomes: Incidence of Complications Associated With the Procedure and/or Device.
Description: Medical Outcomes: Incidence of complications associated with the procedure and/or device.
Time Frame: 24 months
Population: The Secondary Outcome Measures were going to be analyzed at the 24 month visit. However, this study was terminated early due to lack of enrollment and no subjects reached the 24 month analysis visit. There is, therefore, no data to summarize for this Secondary Outcome Measure.
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

7. Secondary Outcome: Medical Outcomes: Comparison of Pre-operative Neurological Reflex Evaluations in the Lower Extremities to Post-operative Findings
Description: Medical Outcomes: Comparison of pre-operative neurological Reflex evaluations in the lower extremities to post-operative findings
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

8. Secondary Outcome: Medical Outcomes: Comparison of Pre-operative Neurological Sensory Responses in the Lower Extremities to Post-operative Findings.
Description: Medical Outcomes: Comparison of pre-operative neurological Sensory Responses in the lower extremities to post-operative findings.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

9. Secondary Outcome: Medical Outcomes: Comparison of Pre-operative Neurological Motors Assessments Evaluated by Straight Leg Raise, Femoral Stretch, and Strength Assessments, to Post-operative Findings.
Description: Medical Outcomes: Comparison of pre-operative neurological Motors assessments evaluated by Straight Leg Raise, Femoral Stretch, and Strength assessments, to post-operative findings.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

10. Secondary Outcome: Patient Reported Outcomes: Comparison of Pre-operative Back Pain Scores to Post-operative Levels as Measured by the (Visual Analog Scale (VAS).
Description: Patient Reported Outcomes: Comparison of pre-operative back pain scores to post-operative levels as measured by the (Visual Analog Scale (VAS).
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

11. Secondary Outcome: Patient Reported Outcomes: Oswestry Disability Index Measurements for Comparison of Pre-operative to Post-operative Evaluations.
Description: Patient Reported Outcomes: Oswestry Disability Index measurements for comparison of pre-operative to post-operative evaluations.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

12. Secondary Outcome: Patient Reported Outcomes: Evaluations of Quality of Life (QOL) as Measured by the SF-12.
Description: Patient Reported Outcomes: Evaluations of Quality of Life (QOL) as measured by the SF-12.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

13. Secondary Outcome: Radiographic Outcomes: Fusion Status Evaluated by X-ray and/or CT Assessments.
Description: Radiographic Outcomes: Fusion status evaluated by x-ray and/or CT assessments.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

14. Secondary Outcome: Radiographic Outcomes: Device Placement Status as Evaluated by X-ray and/or CT Imaging.
Description: Radiographic Outcomes: Device placement status as evaluated by x-ray and/or CT imaging.
Time Frame: 24 months
Population: as for outcome 6
Arm/Group | AccuLIF TL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse Event Reporting according to clinicaltrials.gov definitions
Arm/Group | AccuLIF TL
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AccuLIF TL (N=9)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Enterobacter Cloacae Bacteremia (Infections and infestations) | 1 (1)
Pulmonary Eboli and Pleural Effusions Bilaterally (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AccuLIF TL (N=9)
Radiculitis (Nervous system disorders) | 1 (1)
Dural Tear (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
A total of 100 subjects were planned for enrollment. However, this study was terminated early due to lack of enrollment with only 9 enrolled subjects and 6 treated subjects. No subjects reached the 24 month analysis visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02704689/Prot_SAP_000.pdf